CLINICAL TRIAL: NCT04168099
Title: Comparative Study Between the Efficacy of Oral Gemifloxacin and Intravenous Cefotaxime in Treatment of Spontaneous Bacterial Peritonitis
Brief Title: Oral Gemifloxacin Versus Intravenous Cefotaxime in Treatment of Spontaneous Bacterial Peritonitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBP new treatment
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Cefotaxime; Gemifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefotaxime (Experimental): Cefotaxime intravenous
  Interventions: Drug: Cefotaxime
- Gemifloxacin (Active Comparator): Oral Gemifloxacin
  Interventions: Drug: Gemifloxacin

INTERVENTIONS:
Drug: Cefotaxime — Cefotaxime IV
  Other Names: cefotax, claforan
  Arms: Cefotaxime
Drug: Gemifloxacin — Gemifloxacin oral
  Other Names: gemiflox
  Arms: Gemifloxacin

SUMMARY:
oral Gemifloxacin versus intravenous Cefotaxime in treatment of spontaneous bacterial peritonitis

DETAILED DESCRIPTION:
Comparative Study between the Efficacy of oral Gemifloxacin and intravenous Cefotaxime in treatment of spontaneous bacterial peritonitis

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous bacterial peritonitis

Exclusion Criteria:

* secondary peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with resolution of infection | 6 months
  the total number of patients with resolution of infection

CONTACTS AND LOCATIONS:
Overall Officials: Hala Shaaban El Gendy, Msc, Principal Investigator — Tanta University - Faculty of Medicine; Osama El Sayed Negm, Prof., Principal Investigator — Tropical Medicine Dept.-Tanta University - Faculty of Medicine; Sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tropical Medicine Dept.-Tanta University - Faculty of Medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No